CLINICAL TRIAL: NCT04694118
Title: Comparison of the Effectiveness of Walking Back Exercises and Rebound Therapy in Cerebral Palsy Rehabilitation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Istanbul Medipol University Hospital (Other)
Responsible Party: Principal Investigator, ulkuatasoy2017, Msc.physiotherapist, Istanbul Medipol University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 10840098-604.01.01-E.66352
Record Dates: First submitted 2021-01-01; First posted 2021-01-05 (Actual); Last update posted 2021-01-06 (Actual); Status verified 2021-01

CONDITIONS: Cerebral Palsy, Spastic
Keywords: Cerebral palsy,; neurodevelopmental therapy
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Intervention Model Description: randomise controlled clinical trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 15 hemiparetic cerebral palsy,walking back group (Experimental): GMFM I or II degreed 6-15 age range hemiparetic cerebral palsy
  Interventions: Other: rebound therapy
- 15 hemiparetic cerebral palsy,rebound therapy group (Experimental): GMFM I or II degreed 6-15 age range hemiparetic cerebral palsy
  Interventions: Other: rebound therapy

INTERVENTIONS:
Other: rebound therapy — 3 days a week in 12 weeks
  Other Names: walking back exercise

SUMMARY:
Purpose of the study:

To investigate the effect of walking back exercises and rebound therapy on muscle strength, functionality, balance and aerobic capacity in children with CP Implication for rehabilitation:Determining the effects of rehabilitative interventions (back and forth walking exercises and rebound therapy) to be applied in children with CP with objective measurement methods (muscle US, tetrax balance system) and evaluating the effects of the results on functionality and respiratory parameters

DETAILED DESCRIPTION:
Inclusion Criteria:

Being diagnosed with SP To be in the age range of 6-15 years, where effective communication can be provided in evaluation and treatment processes and when walking begins to mature Having adequate communication skills Being on level I or level II according to GMFM No impairment in visual functions in terms of not affecting postural control responses, Children with family consent

Study design:

Application of the evaluation methods specified at the beginning of the study to all 30 patients with CP who were randomly divided into 2 groups.

Re-evaluations were planned 8 weeks after the first evaluation of all cases who were continuing with structured neurodevelopmental treatment programs. In addition to the ongoing structured neurodevelopmental treatment programs; Group 1: 12 weeks / 3 days 20 minutes walking back exercises on normal ground, Group 2: Rebound therapy exercises, which are arranged according to the functional levels of the cases, will be applied in 12 weeks / 3 days for 20 minutes.

ELIGIBILITY:
Inclusion Criteria:

* Being diagnosed with hemiparetic SP To be in the age range of 6-15 years, where effective communication can be provided in evaluation and treatment processes and when walking begins to mature Having adequate communication skills Being on level I or level II according to KMFSS No impairment in visual functions in terms of not affecting postural control responses, Children with family consent

Exclusion Criteria:

* Orthopedic surgery and / or botulinum toxin-A application for the lower extremity in the last 6 months Being at level III, level IV or level V according to KMFSS Severe convulsion situations that cannot be controlled with drugs Presence of a medical condition that prevents participation in the study Congenital malformation conditions accompanying CP

Ages: 6 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2021-01-04 (Actual); Primary Completion 2021-12-15 (Estimated); Study Completion 2021-12-15 (Estimated)

PRIMARY OUTCOMES:
changes in muscle volume | one measurement at the beginning of the study, second measurement 8 weeks later, 3rd measurement at 12th week following
  ultrasonic imaging

CONTACTS AND LOCATIONS:
Overall Officials: ulku atasoy, msc.pt, Principal Investigator — PhD student
Locations (2):
- Turkey (Türkiye) (2):
  - Umran medical center, Istanbul, Uskudar
  - Ulku Atasoy, Istanbul, Ümraniye

IPD SHARING:
Plan to Share IPD: Yes
all IPD that underlie results in a publication
Supporting Information: Study Protocol
Time Frame: starting 6 months after publication).
Access Criteria: Users and editors with journal memberships published for pubmed users
URL: https://pubmed.ncbi.nlm.nih.gov/